CLINICAL TRIAL: NCT06175936
Title: The Effect of Laughter Yoga on Nursing Students' Well-Being, Perceived Stress and Academic Self-Efficacy: a Randomised Controlled Study
Brief Title: Effect of Laughter Yoga on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olga Incesu, Dr, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Florence Nightingale Faculty-3
Record Dates: First submitted 2023-11-29; First posted 2023-12-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-09

CONDITIONS: Laughter; Stress; Well-Being, Psychological
Keywords: academic self efficacy; laughter yoga; undergraudate nursing education; well-being; stress
MeSH Terms: conditions — Laughter; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laughter yoga group (Experimental): Laughter yoga will be applied to the intervention group in 6 sessions (45 minutes each session). Laughter yoga consists of four parts. Firstly, it starts with warm-up exercises including hand clapping (applause), singing "ho ho ha ha" to relax the facial muscles of the participants and body movements. Secondly, the lungs are prepared with breathing exercises and the mind is prepared for laughter with childish games. This is followed by laughter exercises. Deep breathing exercises are performed between laughter exercises. Laughter yoga is concluded with clapping, singing and relaxation exercises.
  Interventions: Other: Laugther Yoga
- Control group (No Intervention): No laughter yoga intervention will be applied to the control group.

INTERVENTIONS:
Other: Laugther Yoga — Laughter yoga will be applied to the intervention group in 6 sessions (45 minutes each session).
  Arms: Laughter yoga group

SUMMARY:
Nursing students experience different levels of stress due to many reasons such as lifestyle, health, academic performance, competition, choice of profession, new living environment, relationships with peer group and expectations of parents. It is important to develop different coping behaviours/strategies to manage stressful situations. Laughter yoga has proven positive effects on physical and mental health.

The aim of this randomised controlled trial was to examine the effects of laughter yoga on well-being, perceived stress and academic self-efficacy of nursing students.

DETAILED DESCRIPTION:
Laughter yoga, which is a combination of laughter and yoga with breathing techniques, is among traditional and complementary medicine practices. Based on the view that the brain cannot distinguish between real and unreal laughter, laughter yoga aims to benefit from the mental and physical benefits of laughter. Laughter yoga has benefits such as reducing stress and depression symptoms, relaxing muscle tone, increasing blood circulation, lowering blood pressure, increasing melatonin and growth hormone release, increasing pain threshold, strengthening the immune system.

Laughter yoga will be applied to the intervention group in 6 sessions (45 minutes each session). Well-being, Perceived Stress and Academic Self-Efficacy levels of the students will be evaluated before and after the intervention.

Hypotheses of the study; H1: The well-being level of the intervention group increases after laughter yoga.

H2: The academic self-efficacy level of the intervention group increases after laughter yoga.

H3: Perceived stress level of the intervention group decreases after laughter yoga.

H4: The well-being level of the intervention group after laughter yoga is higher than the control group.

H5: The perceived stress level of the intervention group after laughter yoga is lower than the control group.

H6: The academic self-efficacy level of the intervention group after laughter yoga is higher than the control group.

ELIGIBILITY:
Inclusion Criteria:

* To be a 4th year nursing student,
* Volunteer to participate

Exclusion Criteria:

* To take part in the intern programme,
* Simultaneous participation in any methods of complementary medicine,
* Having undergone surgery within the last three months,
* Having a diagnosis of hernia (hernia)
* Having a diagnosis of epilepsy
* Uncontrolled diabetes and cardiovascular disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Well being | 2 weeks post intervention
  The WHO-5 well-being Scale point of the intervention group change laughter yoga.
Academic self-efficcay | 2 weeks post intervention
  The academic self-efficacy point of the intervention group change after laughter yoga.
Stress | 2 weeks post intervention
  The perceived stress scale point of the intervention group change after laughter yoga.

SECONDARY OUTCOMES:
Well being | 2 weeks post intervention
  The WHO-5 well-being Scale point of the intervention group incresad after laughter yoga.
Academic self-efficacy | 2 weeks post intervention
  Academic self-efficacy Scale point of the intervention group incresad after laughter yoga.
Stress | 2 weeks post intervention
  The perceived stress scale point of the intervention group decreased after laughter yoga.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Altıner Yaş, Dr, Study Director — Dr
Locations (1):
- Olga İncesu, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yas MA, Incesu O. The effect of laughter yoga on well-being, perceived stress, and academic self-efficacy in nursing students: A randomized controlled trial. Appl Psychol Health Well Being. 2025 Feb;17(1):e12610. doi: 10.1111/aphw.12610. Epub 2024 Oct 16. PMID 39415513